CLINICAL TRIAL: NCT05700409
Title: Evaluating a Telemedicine-based Intensive Treatment Program for Children and Adolescents With Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Gal Raz-Dubnov MD, MSc, Director, Pediatric LIfestyle Clinic, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC-21-8876
Record Dates: First submitted 2023-01-08; First posted 2023-01-26 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Experimental): The telemedicine arm will include 30, mostly video, consultations for each participant: 3 physician appointments, 7 exercise consultations by our exercise physiologist, 10 dietary consultations by our pediatric dietitian, and 10 psychologist consultations to assist with goal setting and overall well-being. Three visits will be conducted in-office, for physician assessment, smartphone technical assistance and physical measurements (baseline, at 3 months and at the end of the 6-month period). Participants randomized to the telemedicine arm will have a step-counting rewarding app installed on their smartphone by our staff.
  Interventions: Behavioral: Intensive lifestyle consultations
- On-site (Active Comparator): The on-site arm will have 6 monthly visits during the study period, with two consultations performed in each visit - one by the physician or exercise physiologist, and one by our pediatric dietitian.
  Interventions: Behavioral: Intensive lifestyle consultations

INTERVENTIONS:
Behavioral: Intensive lifestyle consultations — detailed above

SUMMARY:
The study objective is to evaluate whether a novel telemedicine-based intensive treatment program for children with obesity is superior to standard on-site care. This will be a randomized, non-blinded (due to the nature of the intervention) study, where 100 children and adolescents aged 10-18 years with obesity will be divided in a 1:1 ratio to either telemedicine or on-site treatments for 6 months.

The telemedicine arm will include 30, mostly video, consultations for each participant: 3 physician appointments, 7 exercise consultations by our exercise physiologist, 10 dietary consultations by our pediatric dietitian, and 10 psychologist consultations to assist with goal setting and overall well-being. Three visits will be conducted in-office, for physician assessment, smartphone technical assistance and physical measurements (baseline, at 3 months and at the end of the 6-month period). Participants randomized to the telemedicine arm will have a step-counting rewarding app installed on their smartphone by our staff.

The in-office arm will have 6 monthly visits during the study period, with two consultations performed in each visit - one by the physician or exercise physiologist, and one by our pediatric dietitian.

The main outcome of the study is BMI standard deviation (z-score) changes, which will be evaluated after 3 and 6 months of treatment during physical office visits in both study arms.

Secondary outcomes will be:

* Body-fat percent changes, assessed by bioimpedance analysis in physical clinic visits.
* Daily step counts, measured by smartphone data/ wearable activity tracker, if available.
* Weight-related quality of life
* Retention and visit cancellation rates.
* Satisfaction of both parent and child from their allocated treatment.

ELIGIBILITY:
Inclusion Criteria:

* Obesity, defined as a BMI at or above 2 standard deviations SDs according to the WHO growth reference
* Owning a smartphone, needed for video conversations, step counting and the gamification app
* Parent consent and child's assent to participate in the program

Exclusion Criteria:

* Significant physical or mental barriers to physical activity and/or to dietary changes (such as autistic spectrum disorder that precludes dietary changes or sufficient exercise, as assessed by the PI)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Participants will decide if they are randomized based on the sub-group of males or of females
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight status | From baseline to 3 months
  BMI z-score change
Weight status | From baseline to 6 months
  BMI z-score change

SECONDARY OUTCOMES:
Body-fat percent changes | From baseline to 3 months
Body-fat percent changes | From baseline to 6 months
Daily step counts | At 3 months
Daily step counts | At 6 months
Weight-related quality of life | Basline
  Scores on the Impact of Weight on Quality of Life (IWQOL)-Kids questionnaire OR "Sizing me up" questionnaire
Weight-related quality of life | 3 months
  Scores on the Impact of Weight on Quality of Life (IWQOL)-Kids questionnaire OR "Sizing me up" questionnaire
Weight-related quality of life | 6 months
  Scores on the Impact of Weight on Quality of Life (IWQOL)-Kids questionnaire OR "Sizing me up" questionnaire
Visit cancellation rates | 6 months
Retention in program | 6 months
  Duration of participation in the program
Satisfaction of allocated treatment | 6 months
  Generic PROM questionnaire used in our hopital

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, State/Province, Israel

IPD SHARING:
Plan to Share IPD: No